CLINICAL TRIAL: NCT02774460
Title: The Precision Hypertension Care Study
Acronym: PHYSIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHY201501
Record Dates: First submitted 2016-03-30; First posted 2016-05-17 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Lisinopril; candesartan cilexetil; candesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Zestril® (Lisinopril) (Active Comparator): Inhibition of angiotensin converting enzyme (ACE inhibitor). Treatment step up: 1-2 weeks (10 mg tablet) Target dose: 5-7 weeks (20 mg tablet)
  Interventions: Drug: Zestril®
- Atacand® (Candesartan) (Active Comparator): Angiotensin receptor blocker. Treatment step up: 1-2 weeks (8 mg tablet) Target dose: 5-7 weeks (16 mg tablet)
  Interventions: Drug: Atacand®
- Norvasc® (Amlodipine) (Active Comparator): Calcium channel blocker. Treatment step up: 1-2 weeks (5 mg tablet) Target dose: 5-7 weeks (10 mg tablet)
  Interventions: Drug: Norvasc®
- Hydrochlorothiazide® (Hydrochlorothiazide) (Active Comparator): Diuretic agent. Treatment step up: 1-2 weeks (12,5 mg tablet) Target dose: 5-7 weeks (25 mg tablet)
  Interventions: Drug: Hydrochlorthiazide®
- Repeated treatment X (Active Comparator): Each patient receives all four treatments, and in addition repeats two of the treatments, labeled X and Y.
  The repeated arms will be given with the same duration and dosing as the other arms.
  Interventions: Drug: Treatment X
- Repeated treatment Y (Active Comparator): Each patient receives all four treatments, and in addition repeats two of the treatments, labeled X and Y.
  The repeated arms will be given with the same duration and dosing as the other arms.
  Interventions: Drug: Treatment Y
- Placebo (Placebo Comparator): This is an unblinded placebo run-in which we use to generate baseline values. Each patient will initiate their participation with these 2 weeks of placebo treatment, taking 1 capsule daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zestril® — Treatment step up: 1-2 weeks (10 mg tablet) Target dose: 5-7 weeks (20 mg tablet)
  Other Names: Lisinopril
  Arms: Zestril® (Lisinopril)
Drug: Atacand® — Treatment step up: 1-2 weeks (8 mg tablet) Target dose: 5-7 weeks (16 mg tablet)
  Other Names: Candesartan
  Arms: Atacand® (Candesartan)
Drug: Norvasc® — Treatment step up: 1-2 weeks (5 mg tablet) Target dose: 5-7 weeks (10 mg tablet)
  Other Names: Amlodipine
  Arms: Norvasc® (Amlodipine)
Drug: Hydrochlorthiazide® — Treatment step up: 1-2 weeks (12,5 mg tablet) Target dose: 5-7 weeks (25 mg tablet)
  Other Names: Hydrochlorthiazide
  Arms: Hydrochlorothiazide® (Hydrochlorothiazide)
Drug: Treatment X — Each patient receives all four treatments, and in addition repeats two of the treatments, labeled X and Y. The repeated arms will be given with the same duration and dosing as the other arms.
  Arms: Repeated treatment X
Drug: Treatment Y — Each patient receives all four treatments, and in addition repeats two of the treatments, labeled X and Y. The repeated arms will be given with the same duration and dosing as the other arms.
  Arms: Repeated treatment Y
Drug: Placebo — This is an unblinded placebo run-in which we use to generate baseline values. Each patient will initiate their participation with these 2 weeks of placebo treatment, taking 1 capsule daily.
  Arms: Placebo

SUMMARY:
The PHYSIC study aims to investigate the potential for precision medicine in the treatment of high blood pressure.

It is a double-blind, randomized, repeated cross-over trial with six treatment periods: four classes of blood pressure-lowering drugs where treatment with two classes are repeated for each patient. The classes of blood pressure-lowering drugs to be tested are a diuretic, a calcium channel blocker, an ACE-inhibitor and an angiotensin receptor blocker.

DETAILED DESCRIPTION:
It is unknown if there is a clinically relevant between-person difference in blood pressure response to a given drug, i.e. if there are responders and non-responders to the drug. If there is no major between-person variation in blood pressure response or side effects of a drug, then there is no potential for precision medicine. It is also unknown if between- person differences in blood pressure response are different for different drugs, and magnitudes of within- and between-person variations in side effects are particularly unknown. Resolving these issues are imperative for the possibilities of precision blood pressure-lowering treatment, and this study aims to initially answer those questions.

If this study proves that there is potential for personalized blood pressure-lowering treatment, investigators will explore the most promising predictors of blood pressure and side effect response to the four major first-line classes of blood pressure-lowering drugs, using several modalities of -omics methods in combination with clinical data. Using these data, investigators will develop and evaluate a point-of-care biomarker panel which will rank the suitability of each of the blood pressure-lowering drug classes for the individual patient in terms of both anticipated blood pressure effect and side effects, thereby providing a suggestion of the priority of the drugs.

The PHYSIC study is a double-blind, randomized, repeated cross-over trial with six treatment periods: four classes of blood pressure-lowering drugs where treatment with two classes are repeated for each patient. The classes of blood pressure-lowering drugs to be tested are a diuretic, a calcium channel blocker, an ACE-inhibitor and an angiotensin receptor blocker. The repeated treatment periods allow investigators to assess whether there is consistent preference of one treatment over another within a blinded patient under different treatment periods. This is a key but often overlooked element in the exploration of the potential for precision medicine.

Evidence-based titration and target doses have been chosen for all four drug classes included. The suggested treatment duration of 7-9 weeks per treatment arm is based on recent guidelines. Patients will be assigned a treatment order based on block randomization ensuring that the same number of patients will repeat each pair of treatments. The study tests several pre-defined hypotheses, which will not be adjusted for multiple testing. The main outcome variable will be variation in daytime ambulatory systolic blood pressure assessed in a blinded fashion.

The screening visit (visit 1) will occur at least two weeks before randomization (visit 2). At screening, consenting patients are assessed to ensure that they meet eligibility criteria initially. Patients who do not meet these criteria must not be enrolled in the study. Patients who do meet these criteria are allocated an enrolment number. The amount of assessment made at this visit includes consent procedures, weight, height, waist, and hip circumference, physical examination, concomitant medication, blood pressure, and blood sampling for safety assessment and DNA genetics. The patient will fill out two questionnaires covering medical history and beliefs about medicine. In order to be introduced to self-reporting symptoms and quality of life collected in electronic diary and get a baseline measurement patients will be asked to log in to and fill the diary under supervision of study staff.

After the screening visit, the patient stops taking any blood pressure-lowering drugs and starts on an unblinded placebo treatment run-in period of two weeks to establish an untreated baseline to be used for characterization of the study sample. During this placebo run-in patients will have access to the electronic diary for reporting symptoms and quality of life. Patients will also be prompted via sms to fill out this diary at home once during this period.

At visit 2, eligibility criteria will be checked once again. Concomitant medication will be checked and blood pressure measured. Other blood pressure-lowering drugs are not allowed as concomitant medication. Baseline assessments made at this visit includes venous blood sampling (DNA methylation, RNA, proteins and metabolites), capillary blood sampling, safety sampling, pulse wave analysis, initiation of the 24h blood pressure and ECG measurement. The study staff will also collect AE ́s via open question and observations. Furthermore patients will also fill out a validated questionnaire to measure perceived symptoms associated with antihypertensive drugs (PERSYVE).

If all criteria are met, the patient will be randomized to the consecutive randomization number and given the first investigational product (IP). The IP will be taken once daily. Each treatment period will be 7-9 weeks (titration dose 2 weeks + target dose 5-7 weeks) and dosing will take place at home.

The day after visit 2 patients will return the 24 h blood pressure and ECG equipment to the clinic.

Between visit 2 and 3 patients are dosing at home. Throughout the study, patients will have access to an electronic diary for reporting symptoms and quality of life, using a validated questionnaire, PERSYVE (only section 2.1 in questionnaire will be used in this study). Patients will also be prompted via sms to fill out these this questionnaire at home at specific time points - at week 3, week 5 and week 7 of each treatment period.

At visit 3 of each treatment period the patient will come fasting to the clinic for venous blood sampling (DNA methylation, RNA, proteins and metabolites), capillary blood sampling, pulse wave analysis, concomitant medication check, blood pressure measurement, and initiation of the 24h blood pressure and ECG measurement. The study staff will also collect adverse events (AEs) via open question and observations. All AEs will be assessed by the Principal Investigator. Furthermore, patients will also fill out two paper questionnaires; PERSYVE section 2.1 (identical to questionnaire in electronic diary) and a treatment preference rating questionnaire. The patient will return all unused IP to site, except for 1 capsule which will be taken the following day. The study personnel will give the patient the next treatment and the patient will undergo a batch, which starts with a 7- day placebo washout period before the next active drug treatment period starts. Lastly, blood samples are obtained and analyzed for safety parameters at visit 3 in the last treatment period only.

At visit 4 (the Week 8 visit) the 24h blood pressure and ECG measurement will end.

One week after visit 4 in the last treatment period, the patient comes to the clinic for a last visit. During this visit the patient will be asked to do an overall treatment preference rating including all treatment periods. An independent and unblinded study physician will be delegated to break the blind for each completed patient and prescribe the preferred IP for continuous use.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥40 years and ≤75 years
2. Previously diagnosed with hypertension with systolic blood pressure between 140 and 159 mm Hg within five years prior to the start of the trial.
3. Pharmacologically untreated or using blood pressure-lowering monotherapy at Visit 1. No blood pressure-lowering medication taken during the placebo run-in period.
4. Office systolic blood pressure between 140 and 179 mm Hg and diastolic blood pressure at or below 109 mm Hg at Visit 2.
5. Patients must give informed consent to participate in the study.

Exclusion Criteria:

1. Medical history, clinical signs or laboratory results indicating secondary hypertension, including primary aldosteronism or renal artery stenosis
2. Evidence of serious hematological, respiratory immunological, renal, hepatic, gastrointestinal, endocrinological, metabolic, neurologic, malignant, psychiatric or other diseases as revealed by medical history, physical examination and/or laboratory assessments.
3. Active gout
4. Previous or present arterial occlusive diseases such as myocardial infarction (MI), stroke or acute arterial insufficiency (unstable angina pectoris or transient ischemic attacks, (TIA)) or heart failure (NYHA class III or IV, or left ventricular systolic dysfunction irrespectively of function class).
5. Moderate or severe aortic or mitral insufficiency.
6. Renal failure, including hemo-dialysis or kidney transplant/s.
7. Atrial fibrillation in need of rate control.
8. Symptomatic hypotension, defined as weakness or syncope upon rising to an erect position associated with a decrease in systolic blood pressure.
9. Diabetes requiring insulin or oral glucose-lowering drugs.
10. Any history of serious abnormal drug reaction to active or inactive compounds in the study drugs, including angioedema.
11. Any condition associated with poor compliance including alcoholism or drug dependence.
12. Patients who will not comply with the study protocol as judged by the Investigator.
13. Women who are pregnant or lactating or not using appropriate contraception for at least 3 months prior to visit 1. Acceptable contraceptive methods are: combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progesterone-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion and vasectomised partner.
14. Continuous use of concomitant medication that can interfere with study medication, i.e. digitalis glucosides, sotalol, cholestyramine, colestipol, NSAID, lithium, carbamazepine, CYP3A4-inhibitors, CYP3A4-inducers, dantrolene, diuretics, aliskiren, gold, sympathomimetics, tricyclic antidepressants, antipsychotics, anaesthetics and potassium supplements.
15. Clinical laboratory assessment outside normal range at visit 1 and judged clinically significant by the Investigator.
16. Previous randomization in present study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Between-person variation in blood pressure-lowering effects of blood pressure-lowering drugs, measured as variation in daytime (10 a.m. to 8 p.m.) ambulatory systolic blood pressure. | This outcome will be analysed based on measurements on the last day of each treatment period (week 7-9).

SECONDARY OUTCOMES:
Between-person variation in side effects of blood pressure-lowering drugs, as measured with a modified section of a validated questionnaire about adverse effects of antihypertensive drugs (PERSYVE section 2.1) | This outcome will be analysed based on data collected on the next to last day of each treatment period (week 7-9).
The difference in patient treatment preferences between the blood pressure lowering drug classes, as measured with a treatment preference rating questionnaire. | This outcome will be analysed based on data collected on the next to last day of each treatment period (week 7-9).
  The questionnaire consists of five questions covering willingness to pay, treatment preference, safety and motivation.
Overall patient treatment preferences measured with a questionnaire on paper. | This outcome will be measured on the last visit for each patient, i.e. week 56.
  The patient is asked to fill out an overall treatment preference rating on paper. The rating is based on a summary of the patients reported symptoms, treatment preference ratings for all treatment periods and a summary of 24 hour blood pressure measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Sundstrom, Professor, Principal Investigator — Uppsala University, Department of Medical Sciences
Locations (1):
- Uppsala University hospital, Internal medicine research, Oscar II, Uppsala, Sweden

REFERENCES:
- [Background] Sundstrom J, Lind L, Nowrouzi S, Lytsy P, Marttala K, Ekman I, Ohagen P, Ostlund O. The Precision HYpertenSIon Care (PHYSIC) study: a double-blind, randomized, repeated cross-over study. Ups J Med Sci. 2019 Jan;124(1):51-58. doi: 10.1080/03009734.2018.1498958. Epub 2018 Sep 28. PMID 30265168
- [Derived] Sundstrom J, Lind L, Nowrouzi S, Hagstrom E, Held C, Lytsy P, Neal B, Marttala K, Ostlund O. Heterogeneity in Blood Pressure Response to 4 Antihypertensive Drugs: A Randomized Clinical Trial. JAMA. 2023 Apr 11;329(14):1160-1169. doi: 10.1001/jama.2023.3322. PMID 37039792